CLINICAL TRIAL: NCT01937351
Title: Evaluation of the Pantheris Optical Coherence Tomography Imaging Atherectomy System for Use in the Peripheral Vasculature
Brief Title: Evaluation of the Pantheris Atherectomy System
Acronym: VISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P0555
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Atherectomy; Optical Coherence Tomography; Lumivascular
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pantheris Treatment Arm (Experimental): Intervention: Atherectomy using the Pantheris system.
  Interventions: Device: Pantheris System

INTERVENTIONS:
Device: Pantheris System — Atherectomy using directional visualization and imaging as an adjunct to fluoroscopy to aid removal of plaque from diseased lower extremity arteries.

SUMMARY:
A non-randomized, prospective, global clinical trial of the Avinger Pantheris System, an atherectomy device that provides directional visualization and imaging as an adjunct to fluoroscopy to aid removal of plaque in diseased lower extremity arteries.

DETAILED DESCRIPTION:
The trial will enroll up to 173 subjects diagnosed with peripheral arterial disease of the lower extremities at up to 20 sites (up to 3 international sites), including 133 Intention to Treat subjects and up to 2 additional Roll-In subjects at each site (up to 40 Roll-In subjects total). The primary disease must be located in reference vessel diameters ≥ 2.5 mm and ≤ 7.0 mm. Trial success is focused on safety including rates of major adverse events through 6 months as adjudicated by a Clinical Events Committee. Effectiveness will be evaluated using technical success, defined as the percent of target lesions that have a residual diameter stenosis <50% post-treatment with the Pantheris device alone as assessed by Angiographic Core Lab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Subject is a candidate for percutaneous intervention for peripheral arterial disease in the legs;
* Subject is willing and able to give informed consent;
* Documented symptomatic atherosclerotic peripheral arterial disease Rutherford Classification 2-5;
* Reference vessel lumen proximal to target lesion ≥ 2.5 mm and ≤ 7.0 mm in diameter by visual estimation;
* Subject has de novo target lesion(s) with stenosis >70% by visual estimation distal to the profunda femoral artery. No more than 2 lesions may be treated with the Pantheris device;
* Target lesion length ≤ 15 cm (may be two tandem lesions that do not exceed 15cm in total length);
* Subject is capable of meeting requirements and be present at the follow-up clinic visits at 30 days and 6 months;
* At least one patent tibial run-off vessel at baseline.

Inclusion Criteria for the 24-month follow up:

* Completed the 6-month follow-up visit
* Re-consented prior to the 24-month follow-up visit

Exclusion Criteria:

* Subject is pregnant or breast feeding;
* Rutherford Class 0 to 1 (asymptomatic and mild claudication);
* Rutherford Class 6 (critical limb ischemia);
* Moderate to severe calcification of the target lesion;
* Acute ischemia and/or acute thrombosis of the Superficial Femoral Artery (SFA)-Popliteal segment;
* In-stent restenosis within the target lesion;
* Target lesion with any type of stent or graft;
* Target lesion in the iliac artery;
* Target lesion stenosis <70%;
* Subjects with significant (≥70%) occlusive lesions proximal to the target lesion not successfully treated during the index procedure (upstream disease) and prior to treatment of the target lesion;
* Endovascular or surgical procedure performed on the index limb less than or equal to 30 days prior to the index procedure;
* Planned endovascular or surgical procedure 30 days after the index procedure;
* Lesion in the contralateral limb requiring intervention during the index procedure or within 30 days of the index procedure;
* Subjects with active systemic infections whether they are being currently treated or not;
* Subjects on chronic hemodialysis or creatinine level >2.0mg/dL;
* Evidence or history of intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stroke within the past 2 months;
* Evidence or history of aneurysmal target vessel within the past 2 months;
* History of severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days;
* Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated;
* Subjects in whom anti-platelet, anticoagulant, or thrombolytic therapy is contraindicated;
* History of heparin-induced thrombocytopenia (HIT);
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/mm2, known coagulopathy, or International Normalized Ratio (INR) >1.5;
* Any thrombolytic therapy within 2 weeks of the index procedure;
* Any clinical and/or angiographic complication attributed to the use of another device prior to the insertion of the study device into the subject;
* Subjects or their legal guardians who have not or will not sign the Informed Consent;
* Subjects who are unwilling or unable to comply with the follow-up study requirements;
* Participation in any study of an investigational device, medication, biologic or other agent within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gray Bennett, MD, Principal Investigator — Jackson Heart Clinic; Billy Crowder, MD, Principal Investigator — Jackson Heart Clinic; Arne Schwindt, MD, Principal Investigator — Muenster Hospital
Locations (21):
- United States (20):
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Cedars Sinai Medical Center/Cardiovascular Research Foundation of Southern California, West Hollywood, California
  - Medstar Washington Hospital, Washington D.C., District of Columbia
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Alexian Brothers Medical Center, Cardiovascular Associates, Elk Grove Village, Illinois
  - Advocate Christ Hospital and Medical Center, Oak Lawn, Illinois
  - St. Joseph's Hospital, Fort Wayne, Indiana
  - Detroit Medical Center Cardiovascular Institute Harper-Hutzel Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - St. Dominic Hospital, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - St. Peters University Hospital, New Brunswick, New Jersey
  - Hatton Institute for Research and Education, Good Samaritan Hospital - Bethesda North, Cincinnati, Ohio
  - Dayton Heart Center/Good Samaritan Hospital, Dayton, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Methodist Hospital, Memphis, Tennessee
  - Austin Heart, Austin, Texas
- Muenster Hospital, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwindt AG, Bennett JG Jr, Crowder WH, Dohad S, Janzer SF, George JC, Tedder B, Davis TP, Cawich IM, Gammon RS, Muck PE, Pigott JP, Dishmon DA, Lopez LA, Golzar JA, Chamberlin JR, Moulton MJ, Zakir RM, Kaki AK, Fishbein GJ, McDaniel HB, Hezi-Yamit A, Simpson JB, Desai A. Lower Extremity Revascularization Using Optical Coherence Tomography-Guided Directional Atherectomy: Final Results of the EValuatIon of the PantheriS OptIcal COherence Tomography ImagiNg Atherectomy System for Use in the Peripheral Vasculature (VISION) Study. J Endovasc Ther. 2017 Jun;24(3):355-366. doi: 10.1177/1526602817701720. Epub 2017 Apr 10. PMID 28393673

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Cohort: The Primary Cohort consisted of either the 1st subject enrolled after the Roll-In cohort or the 1st subject enrolled if the site did not utilize Roll-In subjects.
  The Primary Cohort was analyzed as two separate sub-cohorts: Intention-to-Treat and Per Protocol. The Intention-to-Treat Cohort includes all subjects that were enrolled. The Per Protocol Cohort includes subjects who were enrolled, and had the Pantheris Catheter or Occlusion Sheath device inserted into the vasculature. To be included in this cohort, the Pantheris Catheter also had to be successfully advanced to the intended target lesion. This cohort is a subset of subjects enrolled into the Intention-to-Treat Cohort.
  The Primary Per Protocol Cohort was the cohort used to determine if the primary endpoints of the VISION Study were met.
- Roll-in Cohort: Atherectomy with Pantheris System: The Roll-In Cohort consists of either the 1st subject or 1st and 2nd subjects treated at each site prior to enrollment of subjects into the Primary Cohort. Roll-Ins were designed to provide the Investigator an opportunity to gain experience with the Pantheris System (Catheter and Optical Coherence Tomography-assisted orientation) for learning curve purposes. Certain sites were exempt from enrolling in the Roll-In Cohort.
Period: Overall Study
Arm/Group | Primary Cohort | Roll-in Cohort
Started (Intention-to-Treat) | 134 | 28
Treated w Study Device (Per Protocol) | 130 | 28
30-Day Follow-up | 128 | 27
6-Month Follow-up | 125 | 26
Completed | 125 | 26
Not Completed | 9 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Death | 1 | 0
Not completed — Not treated w device, per protocol fail | 4 | 0

BASELINE CHARACTERISTICS:
Population: The study consisted of Roll-In Cohort and a Primary Analysis Cohort. Up to 2 Roll-In subjects could be treated at each study site prior to initiation of enrollment in the Primary Analysis Cohort.Roll-In subjects were designed to provide the Investigator an opportunity to gain experience with the Pantheris System for learning curve purposes.
Groups:
- Primary Cohort: The Primary Cohort consisted of either the 1st subject enrolled after the Roll-In cohort or the 1st subject enrolled if the site did not utilize Roll-In subjects.
  The Primary Cohort was analyzed as two separate sub-cohorts: Intention-to-Treat and Per Protocol. The Intention-to-Treat Cohort includes all subjects that were enrolled. The Per Protocol Cohort includes subjects who were enrolled, and had the Pantheris Catheter or Occlusion Sheath device inserted into the vasculature. To be included in this cohort, the Pantheris Catheter also had to be successfully advanced to the intended target lesion. This cohort is a subset of subjects enrolled into the Intention-to Treat-Cohort.
  The Primary Per Protocol Cohort was the cohort used to determine if the primary endpoints of the VISION Study were met.
- Roll-In Cohort: The Roll-In Cohort consists of either the 1st subject or 1st and 2nd subjects treated at each site prior to enrollment of subjects into the Primary Cohort. Roll-Ins were designed to provide the Investigator an opportunity to gain experience with the Pantheris System (Catheter and Optical Coherence Tomography-assisted orientation) for learning curve purposes. Certain sites were exempt from enrolling in the Roll-In Cohort.
- Total: Total of all reporting groups
Arm/Group | Primary Cohort | Roll-In Cohort | Total
Number analyzed (Participants) | 134 | 28 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] — Subject age in years
  years | 67.4 (10.5) | 66.7 (10.5) | 67.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 13 | 71
  Male | 76 | 15 | 91
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 80 | 20 | 100
  African American | 35 | 8 | 43
  Hispanic or Latino | 8 | 0 | 8
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
  Unknown or Unavailable | 9 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 127 | 28 | 155
  Germany | 7 | 0 | 7
Weight [Mean (Standard Deviation); unit: pounds] | 179.5 (43.0) | 199.3 (45.3) | 182.9 (44.0)
Height [Mean (Standard Deviation); unit: inches] | 66.8 (3.8) | 66.5 (4.1) | 66.7 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: The primary safety endpoint is defined as freedom from a composite of major adverse events (MAE) through 6-Month follow-up as adjudicated by an independent Clinical Events Committee (CEC). Individual MAEs include:
  1. Cardiovascular related death
  2. Unplanned, major index limb amputation
  3. Clinically driven target lesion revascularization (TLR)
  4. Myocardial infarction
  5. Device related events:
     1. Clinically significant perforation
     2. Clinically significant dissection
     3. Clinically significant embolus
     4. Pseudoaneurysm
Time Frame: Day 0 through 6 Months
Population: Per Protocol: Four Subjects withdrew, 1 subject died (non-CV related), so N=125 instead of 130.
  Intention-to-Treat: Four subjects who were not treated with Pantheris Catheter were exited from the study after the 30-day visit per protocol. Four subjects withdrew, 1 subject died (non-CV related), so N=125 instead of 134.
Measure: Number; unit: percentage of subjects
Groups:
- Primary Cohort: Per Protocol: The 'Primary Cohort: Per Protocol' includes subjects who were enrolled (excluding Roll-in subjects), and had the Pantheris Catheter or Occlusion Sheath device inserted into the vasculature. To be included in this cohort, the Pantheris Catheter also had to be successfully advanced to the intended target lesion. This cohort is a subset of subjects enrolled into the 'Primary Cohort: Intention-to-Treat'.
- Primary Cohort: Intention-to-Treat: The 'Primary Cohort: Intention-to-Treat' includes all subjects enrolled in the study, excluding Roll-in subjects.
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 125 | 125
percentage of subjects | 82.4 | 82.4

2. Primary Outcome: Primary Effectiveness Endpoint: Technical Success
Description: The primary efficacy endpoint of technical success is defined as the percent of target lesions that have a residual diameter stenosis <50% post the Pantheris device alone, as assessed by an independent Angiographic Core Laboratory.
Time Frame: Day 0
Population: Analyses were performed on 'Primary Cohort: Per Protocol' and 'Primary Cohort: Intention-to-Treat', and results were calculated based on number of lesions that were treated.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
Number analyzed (lesions) | 164 | 168
percentage of lesions | 96.3 | 94.0

3. Secondary Outcome: Secondary Safety Endpoint
Description: Freedom from MAEs as defined above, through 30 days (or hospital discharge, whichever is longer) as adjudicated by an independent CEC.
Time Frame: Day 0 through Day 30
Measure: Number; unit: percentage of subjects
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
percentage of subjects | 93.1 | 93.3

4. Secondary Outcome: Secondary Safety Endpoint
Description: Freedom from procedural emboli, defined as a change in any visualized runoff vessel (other than vasospasm and dissection) at any time during the procedure.
Time Frame: Day 0 through 30 days
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
Percentage of subjects | 97.7 [93.4 to 99.5] | 97.8 [93.6 to 99.5]

5. Secondary Outcome: Secondary Safety Endpoint
Description: Freedom from clinically driven Target Vessel Revascularization (TVR) through 6 months, as adjudicated by an independent CEC.
Time Frame: Day 0 through 6 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 125 | 125
Percentage of subjects | 91.2 [84.8 to 95.5] | 91.2 [84.8 to 95.5]

6. Secondary Outcome: Secondary Effectiveness Endpoint: Procedural Success
Description: Procedural success defined as the percent of target lesions that have residual diameter stenosis < 30% post-Pantheris and any other adjunctive therapy, determined by independent Angiographic Core Laboratory.
Time Frame: Day 0
Population: Intention-to-Treat: Angiograms post-adjunctive treatment were not available for one subject. So N=133 participants analyzed instead of 134.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Number of lesions
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 133
Number analyzed (Number of lesions) | 164 | 167
percentage of lesions | 78.7 | 79.0

7. Secondary Outcome: Secondary Effectiveness Endpoint: ABI
Description: Ankle-Brachial Index (ABI) at 30 days. ABI is the ratio of blood pressure in the lower legs to the blood pressure in the arms. ABI between 0.95 and 1.3 is considered normal (free from significant peripheral artery disease).
Time Frame: Day 30
Population: Per Protocol: Data unknown for 18 subjects. Intention-to-Treat: Data unknown for 18 subjects.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 112 | 116
Index | 0.95 (0.16) | 0.95 (0.16)

8. Secondary Outcome: Secondary Effectiveness Endpoint: Rutherford Classification
Description: Rutherford Classification at 30 days. Rutherford Classification is a commonly used clinical means for describing the degree of peripheral artery disease. Rutherford Classifications range from Class 0: asymptomatic, to Class 6: major tissue loss.
Time Frame: Day 30
Population: Per Protocol: Data unknown for 9 subjects. Intention-to-Treat: Data unknown for 9 subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 121 | 125
Percentage of subjects
  Rutherford Classification: 0 - Asymptomatic | 52.9 | 52.8
  Rutherford Classification: 1 - Mild Claudication | 31.4 | 31.2
  Rutherford Classification: 2 - Moderate Claudication | 10.7 | 10.4
  Rutherford Classification: 3 - Severe Claudication | 4.1 | 4.8
  Rutherford Classification: 4 - Ischemic Rest Pain | 0 | 0
  Rutherford Classification: 5 - Minor Tissue Loss | 0.8 | 0.8
  Rutherford Classification: 6 - Major Tissue Loss | 0 | 0

9. Secondary Outcome: Secondary Effectiveness Endpoint: Quality of Life - 12-Item Short Form Survey (SF-12)
Description: Change in Quality of Life measures between Baseline and 30 days using 12-Item Short Form Survey (SF-12). There are two components of the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each yields scores from 0 (representing the worst possible debilitation) to 100 (representing no reduction in quality of life).
Time Frame: Day 30
Population: Per Protocol: Baseline: Data unknown for 5 subjects. Per Protocol: 30-Day: Data unknown for 10 subjects. Intention-to-Treat: Baseline: Data unknown for 5 subjects. Intention-to-Treat: 30-Day: Data unknown for 10 subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
Score on a scale
  Mean SF-12 Mental Component Score: Baseline: number analyzed (Participants) | 125 | 129
  Mean SF-12 Mental Component Score: Baseline | 50.0 (10.3) | 50.3 (10.3)
  Mean SF-12 Mental Component Score: 30-Day: number analyzed (Participants) | 120 | 124
  Mean SF-12 Mental Component Score: 30-Day | 52.1 (9.3) | 52.4 (9.3)
  Mean SF-12 Physical Component Score: Baseline: number analyzed (Participants) | 125 | 129
  Mean SF-12 Physical Component Score: Baseline | 35.6 (8.7) | 35.5 (8.6)
  Mean SF-12 Physical Component Score: 30-Day: number analyzed (Participants) | 120 | 124
  Mean SF-12 Physical Component Score: 30-Day | 41.5 (10.5) | 41.5 (10.4)

10. Secondary Outcome: Secondary Effectiveness Endpoint: Vascular Quality of Life Questionnaire (VascuQoL)
Description: Change in Quality of Life measures between Baseline and 30 days using Vascular Quality of Life Questionnaire (VascuQoL). The VascuQoL is a disease-specific questionnaire developed to assess chronic limb ischemia. VascuQol uses a seven-point scale, with 1 representing the worst score and 7 representing the best score.
Time Frame: Day 30
Population: Per Protocol: 30-Day: Data unknown for 8 subjects. Intention-to-Treat: 30-Day: Data unknown for 8 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
score on a scale
  Mean VascuQoL Score at Baseline | 4.1 (1.2) | 4.1 (1.2)
  Mean VascuQoL Score at 30 Days: number analyzed (Participants) | 122 | 126
  Mean VascuQoL Score at 30 Days | 5.4 (1.5) | 5.4 (1.5)

11. Secondary Outcome: Secondary Effectiveness Endpoint: ABI
Description: Ankle-Brachial Index (ABI) at 6 months. ABI is the ratio of blood pressure in the lower legs to the blood pressure in the arms. ABI between 0.95 and 1.3 is considered normal (free from significant peripheral artery disease).
Time Frame: 6 Month
Population: Per Protocol: Data unknown for 13 subjects. Intention-to-Treat: Four subjects who were not treated with Pantheris Catheter were exited from the study after the 30-day visit per protocol. Data unknown for remaining 13 subjects.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 117 | 117
Index | 0.85 (0.23) | 0.85 (0.23)

12. Secondary Outcome: Secondary Effectiveness Endpoint: Rutherford Classification
Description: Rutherford Classification at 6 months. Rutherford Classification is a commonly used clinical means for describing the degree of peripheral artery disease. Rutherford Classifications range from Class 0: asymptomatic, to Class 6: major tissue loss.
Time Frame: 6 Month
Population: Per Protocol: Data unknown for 10 subjects. Intention-to-Treat: Four subjects who were not treated with Pantheris Catheter were exited from the study after the 30-day visit per protocol. Data unknown for remaining 10 subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 120 | 120
Percentage of subjects
  Rutherford Classification: 0 - Asymptomatic | 41.7 | 41.7
  Rutherford Classification: 1 - Mild Claudication | 29.2 | 29.2
  Rutherford Classification: 2 - Moderate Claudication | 14.2 | 14.2
  Rutherford Classification: 3 - Severe Claudication | 11.7 | 11.7
  Rutherford Classification: 4 - Ischemic Rest Pain | 1.7 | 1.7
  Rutherford Classification: 5 - Minor Tissue Loss | 1.7 | 1.7
  Rutherford Classification: 6 - Major Tissue Loss | 0 | 0

13. Secondary Outcome: Secondary Effectiveness Endpoint: Quality of Life - 12-Item Short Form Survey (SF-12)
Description: Change in Quality of Life measures between Baseline and 6 Months using 12-Item Short Form Survey (SF-12). There are two components of the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each yields scores from 0 (representing the worst possible debilitation) to 100 (representing no reduction in quality of life).
Time Frame: 6 Month
Population: Per Protocol: Baseline: Data unknown for 5 subjects. Per Protocol: 6-Month: Data unknown for 13 subjects. Intention-to-Treat: Baseline: Data unknown for 5 subjects. Intention-to-Treat: 6-Month: Four subjects who were not treated with Pantheris Catheter were exited from the study after the 30-day visit per protocol. Data unknown for remaining 13 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
score on a scale
  Mean SF-12 Mental Component Score: Baseline: number analyzed (Participants) | 125 | 129
  Mean SF-12 Mental Component Score: Baseline | 50.0 (10.3) | 50.3 (10.3)
  Mean SF-12 Mental Component Score: 6-Month: number analyzed (Participants) | 117 | 117
  Mean SF-12 Mental Component Score: 6-Month | 51.0 (11.0) | 51.0 (11.0)
  Mean SF-12 Physical Component Score: Baseline: number analyzed (Participants) | 125 | 129
  Mean SF-12 Physical Component Score: Baseline | 35.6 (8.7) | 35.5 (8.6)
  Mean SF-12 Physical Component Score: 6-Month: number analyzed (Participants) | 117 | 117
  Mean SF-12 Physical Component Score: 6-Month | 39.3 (9.7) | 39.3 (9.7)

14. Secondary Outcome: Secondary Effectiveness Endpoint: Vascular Quality of Life Questionnaire (VascuQoL)
Description: Change in Quality of Life measures between Baseline and 6 months using Vascular Quality of Life Questionnaire (VascuQoL). The VascuQoL is a disease-specific questionnaire developed to assess chronic limb ischemia. VascuQol uses a seven-point scale, with 1 representing the worst score and 7 representing the best score.
Time Frame: 6 Month
Population: Per Protocol: 6-Month: Data unknown for 13 subjects. Intention-to-Treat: 6-Month: Four subjects who were not treated with Pantheris Catheter were exited from the study after the 30-day visit per protocol. Data unknown for remaining 13 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Cohort: Per Protocol | Primary Cohort: Intention-to-Treat
Number analyzed (Participants) | 130 | 134
score on a scale
  Mean VascuQoL Score at Baseline | 4.1 (1.2) | 4.1 (1.2)
  Mean VascuQoL Score at 6 Months: number analyzed (Participants) | 117 | 117
  Mean VascuQoL Score at 6 Months | 5.0 (1.5) | 5.0 (1.5)

ADVERSE EVENTS:
Time Frame: All subjects between enrollment and 6 month follow-up.
Description: There were three types of events in the study. Major Adverse Event (MAE), Serious Adverse Event (SAE), Adverse Event (AE).
  Collection of event data was reported by the site within 24 hours for MAEs, 10 days for SAEs and collected during routine monitoring visits for all other AEs.
Groups:
- Primary Cohort: Pantheris System
Arm/Group | Primary Cohort
All-Cause Mortality (participants affected / at risk) | 5/134
Serious Adverse Events (participants affected / at risk) | 89/134
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort (N=134)
Clinically Driven Target Lesion Revascularization (Vascular disorders) | 10 (10)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Clinically Driven Target Vessel Revascularization (Vascular disorders) | 2 (2)
Access Site Complication (Surgical and medical procedures) | 3 (3)
Bleeding (other than access site) (Injury, poisoning and procedural complications) | 3 (3)
Hypotension, sustained (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Loss of distal collateral flow (Vascular disorders) | 1 (1)
Pain, new onset or worsening from baseline (Vascular disorders) | 3 (3)
Perforation, NHLBI Type I or II (Surgical and medical procedures) | 1 (1)
Emboli requiring intervention to resolve acutely (Vascular disorders) | 3 (3)
Vessel dissection, Grade C or greater (Vascular disorders) | 3 (3)
Pseudoaneurysm defined as device related disruption of the arterial wall (Vascular disorders) | 2 (2)
Vessel dissection, Grade A or B (Surgical and medical procedures) | 4 (4)
Thrombosis (Vascular disorders) | 1 (1)
Unplanned Limb Amputation (Minor or Non-Target Limb) (Surgical and medical procedures) | 1 (1)
Other, Abrasion/Cellutitis (R) UE (Vascular disorders) | 1 (1)
Other, Acute Bronchitis (General disorders) | 1 (1)
Acute Bronchitis (General disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Acute on Chronic Anemia (Blood and lymphatic system disorders) | 1 (1)
Acute on Chronic Kidney Injury (Renal and urinary disorders) | 1 (1)
Acute on Chronic Systolic Congestive Heart Failure Exacerbation (Cardiac disorders) | 1 (1)
Acute Renal Failure (CR 1.06) (Renal and urinary disorders) | 1 (1)
Altered Mental Status Due to Hypoglycemia (General disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atypical Chest Pain (General disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
BTK PAD RLE (Vascular disorders) | 1 (1)
Burn to Left Heel (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Chest Pain Syndrome of Unknown Etiology (General disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Community Acquired RUL Pneumonia (General disorders) | 1 (1)
Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Diastolic Heart Failure (Cardiac disorders) | 1 (1)
Difficulty Swallowing (General disorders) | 1 (1)
Dyspnea (General disorders) | 1 (1)
Dyspnea on Extertion (General disorders) | 1 (1)
Episodic Atrial Fibrillation (Cardiac disorders) | 1 (1)
Gangrenous Changes to Bilateral Metatarsals (Infections and infestations) | 1 (1)
Head Trauma S/P Substantial Fall (Injury, poisoning and procedural complications) | 1 (1)
Hypertensive Crisis (General disorders) | 1 (1)
Hypoglycemia (General disorders) | 1 (1)
Hypokalemia (General disorders) | 1 (1)
Intermittent Chest Discomfort (General disorders) | 1 (1)
Intervention Of Contralateral Leg (Vascular disorders) | 1 (1)
Left Patella Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Multi-organ Failure (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Non Target Revascularization (Vascular disorders) | 1 (1)
NSTEMI (Cardiac disorders) | 1 (1)
PAD-LSFA (Vascular disorders) | 1 (1)
Pain - Right Upper Chest (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Poor Healing Bilateral TMA Wounds Including Infection and Dehiscence (Infections and infestations) | 1 (1)
Pseudoaneurysm at Non-Index Procedure (Vascular disorders) | 1 (1)
Reperfusion Edema (Vascular disorders) | 1 (1)
Respiratory Failure (Cardiac disorders) | 1 (1)
Right Anterior Tibia Hematoma (Blood and lymphatic system disorders) | 1 (1)
Right Leg Ischemia (Vascular disorders) | 1 (1)
RLE Abscess on Shin (Infections and infestations) | 1 (1)
Septic Schock (Infections and infestations) | 1 (1)
Shortness of Breath Due to Influenza A (General disorders) | 1 (1)
Stenosis Contralateral (Right) Leg (Vascular disorders) | 1 (1)
Stenosis of Left Common Fem Artery Following Procedure (Vascular disorders) | 1 (1)
TIA Before Admission (Surgical and medical procedures) | 1 (1)
Ulcer Right Heel (Skin and subcutaneous tissue disorders) | 1 (1)
Unplanned, Nontarget Limb Intervention (Surgical and medical procedures) | 1 (1)
Urinary Retension (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vomiting (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort (N=22)
Pain, New Onset or Worsening from Baseline (General disorders) | 14 (17)
Access Site Complication (Surgical and medical procedures) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the earliest of (a)publication of results, (b)receipt of notice stating that Study has been terminated or (c)18 months after completion or termination, Institution/Investigator (IN) shall have right to publish information & data collected or produced, provided that drafts are provided to Sponsor (SP) at least 60 days prior to the first submission. SP shall comment within 45 days. IN shall delay publication/presentation to enable SP to secure patent or other proprietary protection.